CLINICAL TRIAL: NCT03788928
Title: Study of Plasma mitDNA in Predicting Pancreatic Necrosis in Acute Pancreatitis
Brief Title: Predicting Pancreatic Necrosis Using mitDNA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Soha Mohammad Nageb, spechialist, Assiut University
Other Study IDs: mitDNA in acute pancreatitis
Record Dates: First submitted 2018-12-25; First posted 2018-12-28 (Actual); Last update posted 2018-12-28 (Actual); Status verified 2018-12

CONDITIONS: Pancreatic Necrosis
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Mitochondrial dna serum using qt_PCR
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: serum mitochondrial DNA — serum mitochondrial DNA will be measured using RT-PCR within first 72 hours of symptoms of acute pancreatitis

SUMMARY:
Multiple predictors have been used for early pancreatic necrosis, prediction, detection, and monitoring. These include clinical score systems and circulating biomarkers. Ranson and APACHE II score systems are widely used albeit complex and time-consuming. Recently, the role of circulating biomarkers . Of these novel biomarkers, only CRP has been used routinely in cases of pancreatic necrosis prediction. Mitochondrial DNA (mtDNA) is an extra chromosomal genome occurring in the mitochondria of eukaryotic cells. High levels of mtDNA suggest the presence of pancreatic necrosis and close observation should be given to avoid the development of SAP and pancreatitis infection.

DETAILED DESCRIPTION:
Acute pancreatitis (AP) is inflammation of the pancreas that can become a fatal disease or lead to severe complications . It is characterized clinically by abdominal pain and by increased pancreatic enzyme levels in the blood or urine. Gallstone migration and alcohol abuse are the two major risk factors for AP in humans . According to the updated Atlanta classification, AP is generally divided into mild, moderate or severe pancreatitis according to the presence or absence of multiple organ failure (MOF) or local or systemic complications . Mild pancreatitis has a good prognosis with rapid recovery. The late consequences of AP include impaired pancreatic exocrine function and glucose tolerance, diabetes and development of chronic pancreatitis . Moderately severe AP is characterized by the presence of transient organ failure, local complications or exacerbation of comorbid disease . About one-third of patients with AP develop severe necrotizing pancreatitis with persistent MOF and a high mortality rate. The main goals in the clinical management of AP are adequate fluid resuscitation and the prevention of MOF . Both genetic and environmental factors affect the development and severity of pancreatitis .

Although the pathogenic mechanisms remain largely unknown, increasing evidence suggests that damage-associated molecular pattern molecules (DAMPs) play a central role in the pathogenesis of AP. DAMPs link local tissue damage to systemic inflammation response syndrome (SIRS), which, if severe or sustained, can lead to subsequent MOF and even death . Most DAMPs are recognized by membrane-bound and cytosolic pattern recognition receptors (PRRs) expressed by both immune and nonimmune cell types. This triggers downstream signaling and manifests as sterile inflammation .

The development of AP involves a complex cascade of events , which start with injury or disruption of the pancreatic acini, which then permits the leakage of active pancreatic enzymes including amylolytic, lipolytic and proteolytic enzymes that destroy local tissues. This results in edema, vascular damage, hemorrhage and cell death . In addition to oxidative stress and calcium overload , hypotension and low acinar pH contribute to these initiation processes. After initial production of active pancreatic enzymes, local cell death and systemic inflammation ensue.

Mitochondria, the energy factories of cells, regulate pancreatic cell death through control of the production of adenosine triphosphate (ATP) and reactive oxygen species (ROS), as well as calcium . Dysfunction of mitochondrial calcium uptake and efflux, including elevation of cytosolic calcium from the endoplasmic reticulum, can cause mitochondrial calcium overload, which leads to enhanced generation of mitochondrial ROS and mitochondrial membrane permeabilization. Mitochondria dysfunction-mediated oxidative injury results in endoplasmic reticulum stress, lysosomal damage and the release of proteases (for example, cathepsin and trypsin) to degrade cytosolic proteins that cause pancreatic acinar cell death . Dead, dying and injured pancreatic acinar cells release intra-cellular contents, including DAMPs (for example, high mobility group box 1 [HMGB1], DNA, histones and ATP), which in turn promote infiltration of various immune cells (for example, neutrophils, monocytes and macrophages) and activation of inflammatory signaling pathways.

The severity of experimental AP correlates with the extent and type of cell injury and death. Although multiple forms of cell death exist in physiological and pathological conditions , necrosis and apoptosis are the most widely studied types in both clinical and experimental AP . Necrotic cells are capable of activating proinflammatory and immunostimulatory responses by releasing DAMPs and other molecules, whereas apoptosis is usually considered immunologically silent because the cytoplasmic content is packaged in apoptotic bodies and these membrane-bound cell fragments are rapidly taken up and degraded by phagocytes or autophagy .

Why is the immune system so concerned with cell death? The current notion is that DAMPs released or exposed from dying or dead cells contribute to inflammatory and immune responses to remove dead cells and initiate tissue healing . Failure of this control mechanism can lead to uncontrolled inflammation and serious diseases such as sepsis, arthritis, atherosclerosis, lupus and cancer.

Mitochondria are now recognized not only as central players in cell death but also as an important source of DAMPs. mit-DAMPs, including mitDNA, N-formyl peptides, transcription factor A (TFAM, a mitochondrial HMGB1 homologue) and ROS, play emerging roles in inflammation by the activation of neutrophils, monocytes and macrophages .

The clinical course of AP is generally mild; however, nearly 25% of patients progress into severeAP (SAP) which consists of organ failure and/or pancreatic necrosis (PNec) . Although advances in the diagnosis and management have been made, AP remains a major healthissue to the society, PNec is a major complication of AP which manifests as non-opacified parenchyma with intravenous contrast, as identified via contrast-enhanced CT (CECT) scan. Patients with PNec are more likely to develop pancreatic infection and suffer a greater risk for mortality . Currently,CECT scans remain the "gold standard" to diagnosis PNec clinically . However, the extent of PNec is best seen about 3 days after the presentation of disease and may be missed in early CT scan. In addition, repeated CT scanningis not convenient to monitor changes in necrosis, most not ably for those who are receiving mechanical ventilation or hemofiltration.

Multiple predictors have alternatively been used for early PNec prediction, detection, and monitoring. These include clinical score systems and circulating biomarkers. Ranson and APACHE II score systems are widely used albeit complex and time-consuming. Recently, the role of circulating biomarkers, such as peak creatinine levels, C-reactive protein(CRP), and leptin, has been investigated . Of these novel biomarkers, only CRP has been used routinely in casesof PNec prediction. It is reported that CRP levels higher than 150 mg/l were 86% sensitive, but only 46% specific for pancreatic necrosis . Thus, additional investigationof these novel biomarkers is necessary to further improve PNec prediction.

Mitochondrial DNA (mtDNA) is an extrachromosomal genome occurring in the mitochondria of eukaryotic cells.

Normally, it is strictly contained in mitochondria and notexposed to the innate immune system even following cellapoptosis. However, in times of cell death elicited bystress (e.g., trauma and sepsis), mtDNA is released into systemic circulation and leads to an array of inflammatory reactions . Elevated mtDNA levels have been reported in a variety of clinical situations, including trauma,severe sepsis , and cancer . As PNec is caused by intracellular activation of digestive enzymes and autodigestion.

New therapeutic methods targeting PNec such as endoscopic ultrasound guided transmural drainage and necrosectomy are being tested. Early identification of PNec will be helpful for early treatment. High levels of mtDNA suggest the presence of PNec and close observation should be given to avoid the developmentof SAP and pancreatitis infection.

Necrotic substances released into the blood stimulate the production of inflammatory cytokines and mediators, trigger an inflammatory cascade and eventually lead to the SIRS or multiple organ dysfunction syndrome.

ELIGIBILITY:
Inclusion Criteria:

* all patients diagnosed as acute pancreatitis using elevated serum amylase and contrast enhanced CT scan.

Exclusion Criteria:

* Alchoholics
* Renal impairment

Ages: 16 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be enrolled from Raghi hospital ,Assiut university who will be diagnosed with acute pancreatitis
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
level of serum mitochondrial DNA | baseline
  level of serum mitochondrial DNA in severe acute pancreatitis

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wu L, Xu W, Wang F, Lv T, Yin Z, Song Y. Plasma mtDNA Analysis Aids in Predicting Pancreatic Necrosis in Acute Pancreatitis Patients: A Pilot Study. Dig Dis Sci. 2018 Nov;63(11):2975-2982. doi: 10.1007/s10620-018-5227-9. Epub 2018 Aug 9. PMID 30094625